CLINICAL TRIAL: NCT05911230
Title: Advanced Diffusion MRI to Differentiate Tumor Recurrence From Pseudoprogression in Patients With Glioblastoma and Brain Metastases- AiD GLIO Pilot Trial
Brief Title: Advanced Diffusion MRI to Differentiate Tumor Recurrence From Pseudoprogression in Patients With Glioblastoma and Brain Metastases
Acronym: AiD-GLIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-00888; ko23Cordier
Record Dates: First submitted 2023-06-07; First posted 2023-06-20 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Glioblastoma (GBM)
Keywords: Advanced Diffusion Weighted Magnetic Resonance Imaging (ADW-MRI); Tumor Progress (TP); Pseudo- Progression (PsP)
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: one-arm, monocentric pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ADW-MRI imaging (Other): Patients with a histopathologically proven glioblastoma or brain metastasis who have suspected tumor progression on standard MRI after standard first line therapy and who are candidates for surgical resection and undergoing the ADW-MRI preoperatively.
  Interventions: Diagnostic Test: Advanced diffusion-weighted MRI (ADW-MRI)

INTERVENTIONS:
Diagnostic Test: Advanced diffusion-weighted MRI (ADW-MRI) — An advanced diffusion weighted MRI-sequence will be performed in addition to the routine MRI-diagnostics. This will require the patient to be scanned for additional 30 minutes in a separate MRI-scanner. This technique offers the opportunity of higher sensitivity towards subtle tissue changes associated with increased specificity relating to damage of different tissue components of the CNS. In the case of surgical resection, the histopathological findings will be correlated to the findings of the ADW-MRI.

SUMMARY:
This pilot study investigates whether advanced diffusion-weighted MRI (ADW-MRI) can differentiate between true tumor progression (TP) and a pseudoprogression (PsP) in patients with glioblastoma (GBM) or brain metastases.

DETAILED DESCRIPTION:
Advanced diffusion-weighted MRI (ADW-MRI) offer the opportunity of higher sensitivity towards subtle tissue changes associated with increased specificity relating to damage of different tissue components of the central nervous system (CNS). Within the framework of this study, conventional follow up MRI will be complemented by ADW-MRI in case of suspected tumor recurrence and possible surgical resection of the suspicious tissue. In the case of surgical resection, the histopathological findings will be correlated to the findings of the ADW-MRI. In the depicted pilot phase, the feasibility of the described protocol will be examined and the data concerning correlations between standard histopathologic and genetic workup of the resected tissue and the results concerning tissue features from ADW-MRI will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histopathologically proven glioblastoma or brain metastasis and suspected tumor progress on standard MRI after first line therapy and who are candidates for elective surgical resection.
* Able to give informed consent

Exclusion Criteria:

* Contraindications to MRI (e.g. claustrophobia, pacemaker or other implants without MRI-approval, pregnancy)
* Patients in a life-threatening condition
* Patients in need of emergent surgery
* Histopathological analyses of insufficient quality
* Unable to give informed consent
* Age <18 Years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-24 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Correlation of ADW-MRI-findings to histopathological findings | one time assessment at baseline
  Correlations between standard histopathologic workup of the resected tissue and the results concerning tissue features from ADW-MRI are analyzed (descriptive analysis))

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Cordier, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland